CLINICAL TRIAL: NCT04427280
Title: Cancer: Rapid Diagnostics and Immune Assessment for SARS-CoV-2 (COVID-19)
Acronym: CARDS
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: St George's, University of London (Other); Mologic Ltd (Industry); The Royal Marsden Cancer Charity (Unknown); National Institute for Health Research Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR 5287; 20/NE/0139 (Other: Research Ethics Committee)
Record Dates: First submitted 2020-05-21; First posted 2020-06-11 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Infectious Disease; Cancer; Coronavirus Infection
Keywords: COVID-19; SARS-CoV-2; Cancer; Coronavirus infection
MeSH Terms: conditions — Communicable Diseases; Neoplasms; Coronavirus Infections; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Suspected acute COVID-19 infection
  Interventions: Diagnostic Test: Throat/nose swabs; Diagnostic Test: Saliva collection; Diagnostic Test: Blood collection
- Arm B: Asymptomatic patients with no clinical suspicion of COVID-19
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Diagnostic Test: Throat/nose swabs — Throat/nose swabs will initially be collected at baseline (D0) as part of the diagnostic workup for SARS-CoV-2 infection. Subsequent throat/nose swabs will be taken at D7 (if an inpatient), D14, D28, D42 and D56. Two samples will be taken, one for standard of care testing and one for lateral flow assay and storage for further analysis later such as quantitative PCR.
  Groups: Arm A
Diagnostic Test: Saliva collection — Saliva will be collected at each study visit, by asking the participant to provide a small amount of saliva (approximately 0.5 millilitres (mL)) will be collected. Saliva will be tested by the lateral flow assay when available and excess material stored.
  Groups: Arm A
Diagnostic Test: Blood collection — Approximately 30mL of blood will be taken at each study visit.

SUMMARY:
People with cancer may be at higher risk of poor outcomes with COVID-19 infection. This observational study aims to describe the clinical course of COVID-19 infection in people with cancer and evaluate the utility of antibody and antigen tests for COVID-19. The results of this study will inform clinical practice in the management of cancer patients with COVID-19.

DETAILED DESCRIPTION:
Patients with cancer are thought to have a weakened immune system and small observational case series have suggested patients with cancer are at a higher risk of poor outcome from COVID-19. However, the clinical course of COVID-19 infection amongst cancer patients is not known. In addition, it is unclear when it is appropriate for cancer patients who have recovered from COVID-19 infection to resume anti-cancer therapy.

There is unmet need for diagnostic assays for COVID-19 including tests which can rapidly determine whether the virus has been cleared of the COVID-19. Lateral flow assays investigated in this study are rapid and simple diagnostic tools which can assist in timely diagnostics to inform clinical decision making.

This observational study aims to describe the immunological dynamics and clinical course of COVID-19 in cancer patients and evaluate COVID-19 antibody and antigen lateral flow assays.

The information from our study will add significantly to the understanding of COVID-19 diagnostics and will improve the evidence-base for the management of cancer patients. Furthermore, data from this study could inform the timing and treatment for cancer patients who have recovered from COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Suspected COVID-19 infection undergoing diagnostic testing by SARS-CoV-2 Reverse Transcription-Polymerase Chain Reaction (RT-PCR)
* Metastatic or advanced solid organ malignancy, including lymphoma OR Early stage solid organ malignancy having received therapy (radiotherapy, chemotherapy or targeted agents)
* Patient is ≥ 18 years of age.
* Patient can understand the patient information sheet and is able to provide written informed consent.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (greater than or equal to 18 years of age) presenting with suspected COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheela Rao, MD FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Lau DK, Aresu M, Planche T, Tran A, Lazaro-Alcausi R, Duncan J, Kidd S, Cromarty S, Begum R, Rana I, Li S, Suwaidan AA, Monahan I, Clark DJ, Eckersley N, Staines HM, Groppelli E, Krishna S, Mayora-Neto M, Temperton N, Fribbens C, Watkins D, Starling N, Chau I, Cunningham D, Rao S. SARS-CoV-2 Vaccine Immunogenicity in Patients with Gastrointestinal Cancer Receiving Systemic Anti-Cancer Therapy. Oncologist. 2023 Jan 18;28(1):e1-e8. doi: 10.1093/oncolo/oyac230. PMID 36342104

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 163 patients were recruited in the trial: 11 in Arm A and 152 in Arm B. Of the 11 patients recruited to Arm A, only one patient tested positive for COVID-19 (Coronavirus Disease 2019) at baseline and so was eligible for analysis.
Groups:
- Arm A: Suspected acute COVID-19 infection
  Throat/nose swabs: Throat/nose swabs will initially be collected at baseline (D0) as part of the diagnostic workup for SARS-CoV-2 infection. Subsequent throat/nose swabs will be taken at D7 (if an inpatient), D14, D28, D42 and D56. Two samples will be taken, one for standard of care testing and one for lateral flow assay and storage for further analysis later such as quantitative PCR.
  Saliva collection: Saliva will be collected at each study visit, by asking the participant to provide a small amount of saliva (approximately 0.5mL) will be collected. Saliva will be tested by the lateral flow assay when available and excess material stored.
  Blood collection: Approximately 30mL of blood will be taken at each study visit.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 1 | 152
Completed | 1 (Arm A did not complete recruitment and was abandoned due to insufficient numbers of suspected infected patients attending site.) | 150
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: 153 patients were eligible for analysis in the trial: 1 in Arm A and 152 in Arm B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 1 | 152 | 153
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [67 to 67] | 66 [58 to 74] | 67 [58 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 60 | 60
  Male | 1 | 92 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 128 | 129
  Asian | 0 | 10 | 10
  Other | 0 | 6 | 6
  Caribbean | 0 | 3 | 3
  African | 0 | 2 | 2
  Oriental | 0 | 2 | 2
  Mixed race | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 | 152 | 153
Anatomical site of malignancy [Count of Participants; unit: Participants]
  Colorectal | 0 | 80 | 80
  Oesophagogastric | 0 | 38 | 38
  Hepato pancreatic biliary | 0 | 24 | 24
  Other | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients at Each Sample Timepoint With a Positive Detection of Immunoglobulin G (IgG) Specific Antibodies to SARS-CoV-2 (Spike-protein).
Description: Percentage of patients at each sample timepoint (Day 0 (baseline blood collection), Day 28, Day 56, Day 84) with a positive detection of IgG specific antibodies to SARS-CoV-2 (Severe acute respiratory syndrome coronavirus 2) (spike-protein). Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol.
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients who had at least one blood test taken during the study. Patients were included in the analysis at each timepoint if they had available assay results at that timepoint. The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Arm A: Patients with a suspected acute COVID-19 infection.
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 146 | 0
Percentage of patients
  Spike-protein antibodies: Day 0 | 34.9 [27.2 to 43.3] |
  Spike-protein antibodies: Day 28: number analyzed (Participants) | 128 | 0
  Spike-protein antibodies: Day 28 | 38.3 [29.8 to 47.3] |
  Spike-protein antibodies: Day 56: number analyzed (Participants) | 112 | 0
  Spike-protein antibodies: Day 56 | 52.7 [43 to 62.2] |
  Spike-protein antibodies: Day 84: number analyzed (Participants) | 105 | 0
  Spike-protein antibodies: Day 84 | 61.9 [51.9 to 71.2] |

2. Primary Outcome: Percentage of Patients at Each Sample Timepoint With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Nucleocapsid).
Description: Percentage of patients at each sample timepoint (Day 0 (baseline blood collection), Day 28, Day 56, Day 84) with a positive detection of IgG specific antibodies to SARS-CoV-2 (nucleocapsid). Nucleocapsid (anti-N) antibodies were analysed with the Elecsys SARS-CoV-2 assay on a Cobas analyser (Roche). As specified by the manufacturer, values above a cut-off index (COI) ≥ 1.0 were reported as positive.
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 150 | 0
Percentage of patients
  Nucleocapsid antibodies: Day 0 | 14.7 [9.4 to 21.4] |
  Nucleocapsid antibodies: Day 28: number analyzed (Participants) | 129 | 0
  Nucleocapsid antibodies: Day 28 | 14.0 [8.5 to 21.2] |
  Nucleocapsid antibodies: Day 56: number analyzed (Participants) | 112 | 0
  Nucleocapsid antibodies: Day 56 | 16.1 [9.8 to 24.2] |
  Nucleocapsid antibodies: Day 84: number analyzed (Participants) | 105 | 0
  Nucleocapsid antibodies: Day 84 | 14.3 [8.2 to 22.5] |

3. Secondary Outcome: Percentage of Participants at Each Sample Timepoint With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Spike-protein), in Patients Who Received at Least One SARS-CoV-2 Vaccine Dose Prior to Day 0
Description: Percentage of participants at each sample timepoint (Day 0 (baseline blood collection), Day 28, Day 56, Day 84) with a positive detection of IgG specific antibodies to SARS-CoV-2 (spike-protein), in patients who received at least one SARS-CoV-2 vaccine prior to Day 0. Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol.
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients who received a SARS-CoV-2 vaccine prior to the Day 0 (baseline) timepoint and had at least one blood test taken during the study. Patients were included in the analysis at each timepoint if they had available assay results at that timepoint. The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 63 | 0
Percentage of patients
  Spike-protein antibodies: Day 0 | 61.9 [48.8 to 73.9] |
  Spike-protein antibodies: Day 28: number analyzed (Participants) | 53 | 0
  Spike-protein antibodies: Day 28 | 71.7 [57.7 to 83.2] |
  Spike-protein antibodies: Day 56: number analyzed (Participants) | 48 | 0
  Spike-protein antibodies: Day 56 | 81.3 [67.4 to 91.1] |
  Spike-protein antibodies: Day 84: number analyzed (Participants) | 47 | 0
  Spike-protein antibodies: Day 84 | 91.5 [79.6 to 97.6] |

4. Secondary Outcome: Percentage of Participants at Each Sample Timepoint With a Positive Detection of Pseudovirus Neutralisation (1/40 Titre), in Patients Who Received at Least One SARS-CoV-2 Vaccine Dose Prior to Day 0
Description: Percentage of participants at each sample timepoint (Day 0 (baseline blood collection), Day 28, Day 56, Day 84) with a positive detection of pseudovirus neutralisation (1/40 titre), in patients who received at least one SARS-CoV-2 vaccine prior to Day 0. A pseudovirus assay was used to assess the prevalence of positive neutralising antibodies (achieving pVNT50 at 1/40 serum dilution).
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients who received a SARS-CoV-2 vaccine prior to the Day 0 (baseline) timepoint and had at least one blood test taken during the study. Patients were included in the analysis at each timepoint if they had available assay results at that timepoint. The analysis was restricted to Arm B patients, as test results on pseudovirus neutralisation were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 64 | 0
Percentage of patients
  Pseudovirus neutralisation (1/40 titre): Day 0 | 59.4 [46.4 to 71.5] |
  Pseudovirus neutralisation (1/40 titre): Day 28: number analyzed (Participants) | 53 | 0
  Pseudovirus neutralisation (1/40 titre): Day 28 | 67.9 [53.7 to 80.1] |
  Pseudovirus neutralisation (1/40 titre): Day 56: number analyzed (Participants) | 50 | 0
  Pseudovirus neutralisation (1/40 titre): Day 56 | 60 [45.2 to 73.6] |
  Pseudovirus neutralisation (1/40 titre): Day 84: number analyzed (Participants) | 47 | 0
  Pseudovirus neutralisation (1/40 titre): Day 84 | 83 [69.2 to 92.4] |

5. Secondary Outcome: Percentage of Patients at Each Sample Timepoint With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Spike-protein), in Patients Who Did Not Receive a SARS-CoV-2 Vaccine Dose During the Study.
Description: Percentage of patients at each sample timepoint (Day 0 (baseline), Day 28, Day 56, Day 84) with a positive detection of IgG specific antibodies to SARS-CoV-2 (spike-protein), in patients who did not receive a SARS-CoV-2 vaccine during the study. Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol.
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients who did not receive a SARS-CoV-2 vaccine during the study. Patients were included in the analysis at each timepoint if they had available assay results at that timepoint. The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 49 | 0
Percentage of patients
  Spike-protein antibodies: Day 0 | 8.2 [2.3 to 19.6] |
  Spike-protein antibodies: Day 28: number analyzed (Participants) | 43 | 0
  Spike-protein antibodies: Day 28 | 7 [1.5 to 19.1] |
  Spike-protein antibodies: Day 56: number analyzed (Participants) | 34 | 0
  Spike-protein antibodies: Day 56 | 14.7 [5 to 31.1] |
  Spike-protein antibodies: Day 84: number analyzed (Participants) | 27 | 0
  Spike-protein antibodies: Day 84 | 3.7 [0 to 19] |

6. Secondary Outcome: Percentage of Patients at Each Sample Timepoint With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Nucleocapsid), in Patients Who Did Not Receive a SARS-CoV-2 Vaccine Dose During the Study.
Description: Percentage of patients at each sample timepoint (Day 0 (baseline blood collection), Day 28, Day 56, Day 84) with a positive detection of IgG specific antibodies to SARS-CoV-2 (nucleocapsid), in patients who did not receive a COVID-19 vaccine during the study. Nucleocapsid (anti-N) antibodies were analysed with the Elecsys SARS-CoV-2 assay on a Cobas analyser (Roche). As specified by the manufacturer, values above a cut-off index (COI) ≥ 1.0 were reported as positive.
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients who did not receive any SARS-CoV-2 vaccine prior to the Day 0 (baseline) timepoint, had at least one blood test taken during the study, and did not receive a SARS-CoV-2 vaccine during the study. Patients were included in the analysis at each timepoint if they had available assay results at that timepoint. The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 51 | 0
Percentage of patients
  Nucleocapsid antibodies: Day 0 | 7.8 [2.2 to 18.9] |
  Nucleocapsid antibodies: Day 28: number analyzed (Participants) | 44 | 0
  Nucleocapsid antibodies: Day 28 | 6.8 [1.4 to 18.7] |
  Nucleocapsid antibodies: Day 56: number analyzed (Participants) | 34 | 0
  Nucleocapsid antibodies: Day 56 | 11.8 [3.3 to 27.5] |
  Nucleocapsid antibodies: Day 84: number analyzed (Participants) | 27 | 0
  Nucleocapsid antibodies: Day 84 | 3.7 [0 to 19] |

7. Secondary Outcome: Percentage of Participants With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Spike-protein), at Time Periods Relative to the Date of 1st SARS-CoV-2 Vaccine Dose
Description: Percentage of participants with a positive detection of IgG specific antibodies to SARS-CoV-2 (spike-protein), at time periods relative to the date of 1st SARS-CoV-2 vaccine dose. Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol.
Time Frame: 0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days from the date of the patient's 1st SARS-CoV-2 vaccine dose (relative to each patient)
Population: Patients who received a SARS-CoV-2 vaccine prior to the Day 0 (baseline) timepoint and had at least one blood test taken during the study. Patients were analysed if they had available assay results during at least one of the following time periods from the date of their 1st vaccine dose (0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days). The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 57 | 0
Percentage of patients
  Spike-protein antibodies: 0-19 days: number analyzed (Participants) | 50 | 0
  Spike-protein antibodies: 0-19 days | 30 [17.9 to 44.6] |
  Spike-protein antibodies: 20-39 days | 70.2 [56.6 to 81.6] |
  Spike-protein antibodies: 40-59 days: number analyzed (Participants) | 45 | 0
  Spike-protein antibodies: 40-59 days | 64.4 [48.8 to 78.1] |
  Spike-protein antibodies: 60-79 days: number analyzed (Participants) | 39 | 0
  Spike-protein antibodies: 60-79 days | 79.5 [63.5 to 90.7] |
  Spike-protein antibodies: 80-99 days: number analyzed (Participants) | 43 | 0
  Spike-protein antibodies: 80-99 days | 86.1 [72.1 to 94.7] |

8. Secondary Outcome: Percentage of Participants With a Positive Detection of Pseudovirus Neutralisation, at Time Periods Relative to the Date of 1st SARS-CoV-2 Vaccine Dose
Description: Percentage of participants with a positive detection of pseudovirus neutralisation (1/40 titre), at time periods relative to the date of 1st SARS-CoV-2 vaccine dose. A pseudovirus assay was used to assess the prevalence of positive neutralising antibodies (achieving pVNT50 at 1/40 serum dilution)
Time Frame: as for outcome 7
Population: Patients who received a SARS-CoV-2 vaccine prior to the Day 0 (baseline) timepoint and had at least one blood test taken during the study. Patients were analysed if they had available assay results during at least one of the following time periods from the date of their 1st vaccine dose (0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days). The analysis was restricted to Arm B patients, as pseudovirus neutralisation test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 57 | 0
Percentage of patients
  Pseudovirus neutralisation (1/40 titre): 0-19 days: number analyzed (Participants) | 52 | 0
  Pseudovirus neutralisation (1/40 titre): 0-19 days | 40.4 [27 to 54.9] |
  Pseudovirus neutralisation (1/40 titre): 20-39 days | 71.9 [58.5 to 83] |
  Pseudovirus neutralisation (1/40 titre): 40-59 days: number analyzed (Participants) | 45 | 0
  Pseudovirus neutralisation (1/40 titre): 40-59 days | 57.8 [42.2 to 72.3] |
  Pseudovirus neutralisation (1/40 titre): 60-79 days: number analyzed (Participants) | 40 | 0
  Pseudovirus neutralisation (1/40 titre): 60-79 days | 65 [48.3 to 79.4] |
  Pseudovirus neutralisation (1/40 titre): 80-99 days: number analyzed (Participants) | 44 | 0
  Pseudovirus neutralisation (1/40 titre): 80-99 days | 68.2 [52.4 to 81.4] |

9. Secondary Outcome: Sensitivity of the Siemens Test (Spike-protein) at Each Sample Timepoint (D0, D28, D56, D84), Against Pseudovirus Neutralisation Results at the PV50 Threshold.
Description: Sensitivity: the percentage of participants with a positive detection of IgG specific antibodies to SARS-CoV-2 (spike protein) out of those who had a positive neutralisation detection at the PV50 threshold from the pseudovirus assay, at each sample timepoint. Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol. A pseudovirus assay was used to assess the prevalence of positive neutralising antibodies (achieving pVNT50 at 1/40 serum dilution).
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients who had at least one blood test taken during the study. Patients were included in the analysis at each timepoint if they had available assay results at that timepoint. The analysis was restricted to Arm B patients, as antibody and pseudovirus neutralisation test results were not available for the eligible Arm A patient.
Measure: Number; unit: Sensitivity (%)
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 146 | 0
Sensitivity (%)
  Day 0 | 88.5 |
  Day 28: number analyzed (Participants) | 128 | 0
  Day 28 | 80.8 |
  Day 56: number analyzed (Participants) | 112 | 0
  Day 56 | 89.8 |
  Day 84: number analyzed (Participants) | 105 | 0
  Day 84 | 96.7 |

10. Secondary Outcome: Specificity of the Siemens Test (Spike-protein) at Each Sample Timepoint (D0, D28, D56, D84), Against Pseudovirus Neutralisation Results at the PV50 Threshold.
Description: Specificity: the percentage of participants with a negative detection of IgG specific antibodies to SARS-CoV-2 (spike protein) out of those who had a negative neutralisation detection at the PV50 threshold from the pseudovirus assay, at each sample timepoint. Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol. A pseudovirus assay was used to assess the prevalence of positive neutralising antibodies (achieving pVNT50 at 1/40 serum dilution)
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: as for outcome 9
Measure: Number; unit: Specificity (%)
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 146 | 0
Specificity (%)
  Day 0 | 94.7 |
  Day 28: number analyzed (Participants) | 128 | 0
  Day 28 | 90.8 |
  Day 56: number analyzed (Participants) | 112 | 0
  Day 56 | 76.2 |
  Day 84: number analyzed (Participants) | 105 | 0
  Day 84 | 86.4 |

11. Post Hoc Outcome: Percentage of Participants With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Spike-protein), at Time Periods Relative to the Date of 2nd SARS-CoV-2 Vaccine Dose
Description: Percentage of participants with a positive detection of IgG specific antibodies to SARS-CoV-2 (spike-protein), at time periods relative to the date of 2nd vaccine dose (0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days). Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol.
Time Frame: 0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days from the date of the patient's 2nd SARS-CoV-2 vaccine dose (relative to each patient)
Population: Patients who received a second SARS-CoV-2 vaccine, had a vaccine prior to the Day 0 (baseline) timepoint and had at least one blood test taken during the study. Patients were analysed if they had available assay results during at least one of the following time periods from the date of their 2nd vaccine dose (0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days). The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 38 | 0
Percentage of patients
  Spike-protein antibodies: 0-19 days | 84.2 [68.7 to 94] |
  Spike-protein antibodies: 20-39 days: number analyzed (Participants) | 25 | 0
  Spike-protein antibodies: 20-39 days | 96 [79.6 to 99.9] |
  Spike-protein antibodies: 40-59 days: number analyzed (Participants) | 20 | 0
  Spike-protein antibodies: 40-59 days | 95 [75.1 to 99.9] |
  Spike-protein antibodies: 60-79 days: number analyzed (Participants) | 10 | 0
  Spike-protein antibodies: 60-79 days | 100 [NA to NA] — Confidence interval bounds were not defined as the percentage of patients with a positive detection was 100%. |
  Spike-protein antibodies: 80-99 days: number analyzed (Participants) | 5 | 0
  Spike-protein antibodies: 80-99 days | 100 [NA to NA] — Confidence interval bounds were not defined as the percentage of patients with a positive detection was 100%. |

12. Post Hoc Outcome: Percentage of Participants With a Positive Detection of Pseudovirus Neutralisation, at Time Periods Relative to the Date of 2nd SARS-CoV-2 Vaccine Dose
Description: Percentage of participants with a positive detection of pseudovirus neutralisation (1/40 titre), at time periods relative to the date of 2nd SARS-CoV-2 vaccine dose (0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days). A pseudovirus assay was used to assess the prevalence of positive neutralising antibodies (achieving pVNT50 at 1/40 serum dilution)
Time Frame: as for outcome 11
Population: Patients who received a second SARS-CoV-2 vaccine, and had a vaccine prior to the Day 0 (baseline) timepoint. Patients were analysed if they had available assay results during at least one of the following time periods from the date of their 2nd vaccine dose (0-19 days, 20-39 days, 40-59 days, 60-79 days, 80-99 days). The analysis was restricted to Arm B patients, as pseudovirus neutralisation test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 39 | 0
Percentage of patients
  Pseudovirus neutralisation (1/40 titre): 0-19 days | 76.9 [60.7 to 88.9] |
  Pseudovirus neutralisation (1/40 titre): 20-39 days: number analyzed (Participants) | 25 | 0
  Pseudovirus neutralisation (1/40 titre): 20-39 days | 84 [63.9 to 95.5] |
  Pseudovirus neutralisation (1/40 titre): 40-59 days: number analyzed (Participants) | 20 | 0
  Pseudovirus neutralisation (1/40 titre): 40-59 days | 90 [68.3 to 98.8] |
  Pseudovirus neutralisation (1/40 titre): 60-79 days: number analyzed (Participants) | 10 | 0
  Pseudovirus neutralisation (1/40 titre): 60-79 days | 90 [55.5 to 99.7] |
  Pseudovirus neutralisation (1/40 titre): 80-99 days: number analyzed (Participants) | 5 | 0
  Pseudovirus neutralisation (1/40 titre): 80-99 days | 100 [NA to NA] — Confidence interval bounds were not defined as the percentage of patients with a positive detection was 100%. |

13. Primary Outcome: Percentage of Patients at Each Sample Timepoint With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Spike-protein), Across Patients Who Had Blood Test Results Available at All Blood Sample Timepoints (Day 0, Day 28, Day 56, Day 84)
Description: Percentage of patients at each sample timepoint (Day 0 (baseline blood collection), Day 28, Day 56, Day 84) with a positive detection of IgG specific antibodies to SARS-CoV-2 (spike-protein). Serum SARS-CoV-2 S1 RBD Spike antibodies (anti-S) were measured using the COV2T assay on an Atellica analyser (Siemens). Index values ≥ 1.0 were considered positive as per the manufacturer's protocol.
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients were included in the analysis at each timepoint if they had available assay results across all blood sample timepoints (Day 0, Day 28, Day 56, Day 84). The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 78 | 0
Percentage of patients
  Spike-protein antibodies: Day 0 | 34.6 [24.2 to 46.2] |
  Spike-protein antibodies: Day 28 | 41 [30 to 52.7] |
  Spike-protein antibodies: Day 56 | 50 [38.5 to 61.5] |
  Spike-protein antibodies: Day 84 | 60.3 [48.5 to 71.2] |

14. Primary Outcome: Percentage of Patients at Each Sample Timepoint With a Positive Detection of IgG Specific Antibodies to SARS-CoV-2 (Nucleocapsid), Across Patients Who Had Blood Test Results Available at All Blood Sample Timepoints (Day 0, Day 28, Day 56, Day 84)
Description: as for outcome 2
Time Frame: Blood collection timepoints: Day 0 (baseline), Day 28, Day 56, Day 84
Population: Patients were included in the analysis at each timepoint if they had available assay results at all blood sample timepoints (Day 0, Day 28, Day 56, Day 84). The analysis was restricted to Arm B patients, as antibody test results were not available for the eligible Arm A patient.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B | Arm A
Number analyzed (Participants) | 80 | 0
Percentage of patients
  Nucleocapsid antibodies: Day 0 | 12.5 [6.2 to 21.8] |
  Nucleocapsid antibodies: Day 28 | 12.5 [6.2 to 21.8] |
  Nucleocapsid antibodies: Day 56 | 12.5 [6.2 to 21.8] |
  Nucleocapsid antibodies: Day 84 | 12.5 [6.2 to 21.8] |

ADVERSE EVENTS:
Time Frame: Data on adverse events were not recorded for the purposes of this study.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT04427280/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT04427280/SAP_001.pdf
  • Informed Consent Form: Arm A (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT04427280/ICF_002.pdf
  • Informed Consent Form: Arm B (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT04427280/ICF_003.pdf